CLINICAL TRIAL: NCT06544772
Title: Pilot Study of a Smartphone-Based Program in Adults to Measure Switch Rates From Cigarettes to Smoke-free Nicotine Products (C-520)
Brief Title: Study of a Smartphone-Based Switch Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pivot Health Technologies Inc. (Industry)
Responsible Party: Principal Investigator, MacKenzie Utley, Senior Clinical Research Associate, Pivot Health Technologies Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C-520
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; cigarette cessation; digital health; mobile apps
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Pivot cigarette smoking cessation program (Experimental): A commercially available mobile phone app and program for smoking cessation
  Interventions: Device: Pivot cigarette smoking cessation program

INTERVENTIONS:
Device: Pivot cigarette smoking cessation program — The Pivot cigarette smoking cessation program comprises a mobile personal breath carbon monoxide sensor (Pivot Breath Sensor) and a smartphone app (Pivot app) with in-app asynchronous SMS text-based coaching with a certified human tobacco cessation coach.

SUMMARY:
Prospective, open label, single center clinical study enrolling up to 120 participants to evaluate the Pivot cigarette smoking cessation program in adult smokers, previously unable to quit, who also use other smoke-free nicotine product(s) (poly-use) and wish to stop cigarette smoking by switching to these smoke-free nicotine products.

DETAILED DESCRIPTION:
This is a prospective, open label, single center clinical study conducted with Institutional Review Board approval enrolling up to 120 adult participants who report cigarette smoking and concurrent use of smoke-free nicotine product(s), and wish to switch completely off cigarettes. The study will be performed remotely on an ambulatory basis.

Participants will be asked to set up and use the Pivot cigarette smoking cessation program which comprises a mobile personal breath carbon monoxide sensor (Pivot Breath Sensor) and a smartphone app (Pivot app) with in-app asynchronous text-based coaching with a certified human tobacco cessation coach. The study duration is 26 weeks, with main outcomes assessed at 12 weeks (primary endpoint) and 26 weeks. Participants will receive online questionnaires at intervals throughout the study. Participants who indicate abstinence from cigarette smoking at 12 weeks will be invited to do a video call biovalidation visit in which they perform an observed breath sample using their Pivot breath sensor.

Potential participants will complete an online screening form. Eligible participants will be called to confirm eligibility, discuss the study, and have their questions about the study answered. Interested eligible participants will complete the electronic informed consent form and baseline questionnaire prior to downloading the app on their smartphone.

The investigators aim to assess the performance of the Pivot program among adult smokers who also use other smoke-free nicotine products, with a focus on assessing trial feasibility, program acceptability, use and engagement, changes in attitudes towards switching from cigarettes to smoke-free nicotine products and changes in cigarette, nicotine product use, and carbon monoxide (CO) values over the course of the 26-week study, as well as participant feedback on the set-up, design, use experience, and impact of the program.

ELIGIBILITY:
Inclusion Criteria:

* 21-65 years of age
* Smoke ≥ 5 CPD on ≥ 5 days per week
* Have smoked cigarettes for ≥ the last 6 months
* Current use of ≥1 reduced risk smoke-free nicotine product which includes e-cigarettes/vaping, oral nicotine pouch (ONP; ex. Zyn, On, Velo), or heat-not-burn (ex. IQOS, Glo, Ploom, Pulze)
* Planning to quit cigarette smoking by switching to a reduced risk smoke-free nicotine product
* Self-report of ≥ 1 past failed cigarette smoking quit attempt
* Resident of the United States
* Able to read and comprehend English
* Owns and uses a smartphone compatible with the study app (iPhone 6 and above with operating system iOS 15 and above, or, Android 7.0 and above with operating system Android 7.0 and above)
* Has daily internet access on smartphone
* Comfortable downloading and using smartphone apps
* Willing to sign the Informed Consent Form

Exclusion Criteria:

* Pregnant or breast-feeding (self-report)
* Use of other smoking cessation apps, coaching, classes, or quit programs at entry or within previous 30 days
* Current use of nicotine replacement therapy (NRT), chewing tobacco or cigars
* Smokes marijuana ≥ 4 days per week
* Current enrollment in another clinical trial
* Failure to provide contact or collateral information, and/or failure to verify email address
* Participation in a previous study sponsored by Pivot Health Technologies Inc. (formerly Carrot Inc.)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2024-08-16 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-06-09 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who completely switch from cigarettes to a smoke-free nicotine product by 12 weeks | 12 weeks
  The proportion of participants who self-report 7-day point prevalence abstinence (PPA) from cigarettes at 12 weeks and self-report the use of 1 or more smoke-free nicotine products at 12 weeks.

SECONDARY OUTCOMES:
Trial feasibility: online screening form completers | Enrollment
  Trial feasibility in study enrollment is assessed via 3 measures, the first being the proportion of unique (non-duplicate) online screening form completers who are eligible for the screening study phone call.
Trial feasibility: eligible online screening form completers | Enrollment
  Trial feasibility in study enrollment is assessed via 3 measures, the second being the proportion of unique (non-duplicate) online screening form completers who are eligible for the screening study phone call and complete the screening study phone call.
Trial feasibility: study enrollment | Enrollment
  Trial feasibility in study enrollment is assessed via 3 measures, the third being the proportion of unique (non-duplicate) online screening form completers who complete the screening phone call and enroll in the study. Enrollment is defined as completing the HIPAA authorization form and electronic informed consent form (ICF), the online baseline questionnaire, and registration in the Pivot app.
Trial feasibility: Study completion | 12 and 26 weeks
  Trial feasibility in study completion is assessed via one measure:
  1) The proportion of enrolled participants who complete the study questionnaire at 12 weeks, 26 weeks, and both timepoints.
Engagement with program - app openings/sessions | 12 weeks
  Collected via back-end app data collection. Engagement is specifically assessed with number of times the Pivot app was opened (number of app openings/sessions).
Engagement with program - number of days with app openings/sessions | 12 weeks
  Collected via back-end app data collection. Engagement is specifically assessed with the number of days over which the app was opened by participants (at least one app session).
Engagement with program - number of weeks with app openings/sessions | 12 weeks
  Collected via back-end app data collection. Engagement is specifically assessed with the number of weeks over which the app was opened by participants (at least one app session).
Engagement with program - average duration of app sessions | 12 weeks
  Collected via back-end app data collection. Engagement is specifically assessed with the average duration of app sessions completed by participants. Outcome unit of measure = duration in minutes.
Engagement with program - use of app features | 12 weeks
  Collected via back-end app data collection. Engagement is specifically assessed with the use of app features (practice switches, challenges, logging cigarettes) by participants. Reported as the number of times each app feature was used.
Engagement with coaching | 12 weeks
  Collected via back-end app data collection. Engagement is specifically assessed with average number of messages sent by coach to participant per week and average number of messages sent by participant to coach per week.
Average number of weeks with coaching engagement | 12 weeks
  Collected via back-end app data collection. Specifically, the average number of weeks with at least one message sent from participant to coach, and the average number of weeks with at least one message sent from coach to participant.
User satisfaction - Net Promoter Score | 4, 12 and 26 weeks
  Specifically regarding likelihood to recommend to a friend, Net Promoter Score (NPS). Participants asked: "How likely are you to recommend the Pivot program to a friend or colleague?". Answered on a range from 1-10; 1 = Not at all likely, and 10 = Very likely. A higher score indicates greater user satisfaction and promotion of the program.
User feedback - setting up and getting started with the program | 1 week
  Specifically regarding set-up and getting started with the program. Participants asked: "How easy or difficult was it to set-up and get started in the Pivot program?". Answered on a range from 1-10; 1 = Very difficult, and 10 = Very easy. A higher score indicates greater ease of program set-up and getting started.
Participant need for the program | 4 weeks
  Participants are asked: "Which of the following best describes your need for the Pivot program?". Answer choices include the following: "I really need this program", "I somewhat need this program", "I don't need this program", and "I am not at all interested in this program".
User satisfaction - helpful for switching | 8 weeks
  Specifically regarding whether the program was useful in helping participants quit vaping. Participants are asked: "Which of the following best describes the Pivot program's ability to help someone switch off smoking to smoke-free nicotine products?". Answer choices include the following: "The program is extremely helpful to switching"; "The program is helpful to switching"; "The program does not affect being able to switch"; and "The program makes switching harder".
Change in Self-Efficacy | 6, 12 and 26 weeks
  Change in Self-Efficacy from baseline assessment. Self-Efficacy is measured through the 6-item Smoking Abstinence Self-efficacy Questionnaire (SASEQ) (Spek V, et al. Int.J. Behav. Med. (2013) 20:444-449).
  SASEQ score is on a scale of 0-24. Each of the 6 questions is answered on a 5-point Likert scale (0-4). Greater scores indicate greater self-efficacy toward quitting smoking.
Change in Expected Difficulty in Staying Switched | 4, 8 and 12 weeks
  Change in expected difficulty to stay switched from baseline assessment. Participants asked: "How difficult do you think it would be to stay switched?". Participant self-report on scale 1-10 (1=Really hard to stay switched, 10=Really easy to stay switched).
Change in Confidence Levels Towards Switching | 4, 8 and 12 weeks
  Change in confidence levels towards switching from baseline assessment. Participants asked: "If you were to switch from cigarette smoking to a smoke-free nicotine product right now, how successful would you be?". Participant self-report on scale 1-10 (1=Not at all successful, 10=Completely successful).
Desire to Switch (Yes/No) | 4 weeks
  Participants are asked: "Would you like to completely switch from cigarette smoking to a smoke-free nicotine product?". Participants answer "Yes" or "No".
Interest in Switching | Baseline
  Participants are asked: "How interested are you in completely switching from cigarettes to smoke-free nicotine products?". Participants are provided the following answers to choose from: "Extremely", "Somewhat", "Not interested".
Self-Reported Switch | 12 and 26 weeks
  Participant self-report of 7-day and 30-day point prevalence abstinence (PPA) from cigarettes + use of 1 or more smoke-free nicotine products.
Biochemically Confirmed Abstinence | 12 weeks
  Participants who report they have achieved at least 7-day point prevalence abstinence (self-reported switch) at 12 weeks will undergo a videoconference visit with study staff in which they provide a witnessed breath sample using a provided personal mobile carbon monoxide breath sensor. Breath sample values less than 10 ppm (parts per million) will be considered consistent with biochemical abstinence.
Self-Reported Continuous Maintenance of Switch | 26 weeks
  Defined as self-report of 7-day (or greater) PPA from cigarettes at 12 weeks + self-report of 30-day PPA at 26 weeks + use of at least one smoke-free nicotine product at both timepoints.
Duration of Self-Reported Switch | 12 and 26 weeks
  Defined as the duration from present date (date of questionnaire completion) to self-reported date of last cigarette, asked at 12 weeks and 26 weeks, in participants reporting current use of smoke-free nicotine products.
Duration of Abstinence from Cigarettes | 12 and 26 weeks
  Defined as duration from present date (date of questionnaire completion) to self-reported date of last cigarette.
Self-Reported Use/Abstinence of Other Nicotine-Containing Products | 12 and 26 weeks
  Participant self-report of any nicotine products, other than cigarettes, that they currently use.
Duration of Self-Reported Abstinence from All Nicotine Products | 12 and 26 weeks
  Defined as the duration from present date (date of questionnaire completion) to self-reported date of last use of nicotine product, asked at 12 weeks and 26 weeks.
Proportion with ≥ 50% CPD Reduction | 12 and 26 weeks
  Proportion of participants who reduced their cigarettes per day (CPD) by ≥ 50% compared to baseline.
Average % CPD Reduction | 12 and 26 weeks
  The average proportion of reduction in cigarettes per day (CPD) at follow-up compared to baseline.
Change in CPD | 12 and 26 weeks
  The proportion of participants whose change in cigarettes per day (CPD) decreased, increased, or remained unchanged from baseline to follow-up.
Change in Nicotine Product Use | 12 and 26 weeks
  The proportion of participants whose change in nicotine product use decreased, increased, or remained unchanged from baseline to follow-up.
Attempts to Switch | 4, 8, 12 and 26 weeks
  Self-reported number of attempts to switch from cigarettes to smoke-free nicotine products during the study. Participants are asked: "Since you began the study, how many times have you tried to switch from smoking cigarettes to a smoke-free nicotine product where you've gone at least 1 day without smoking a cigarette, even a single puff?".
Attempts to Quit Nicotine Products | 8, 12 and 26 weeks
  Self-reported number of attempts to stop using nicotine products other than cigarettes during the study.
Change in breath CO values for frequent breath sensor users | 1, 4, 8 and 12 weeks
  Change in average weekly breath carbon monoxide (CO) value and average maximum weekly breath CO value in participants with ≥ 4 samples per week (frequent breath sensor users) for the weeks of 1, 4, 8, and 12.
Change in breath CO values on Saturdays | 1-12 weeks
  Change in average Saturday breath carbon monoxide (CO) value over weeks 1-12 in participants with at least one 1 breath sample on the Saturday in question.
Change in participant self-reported health | 26 weeks
  Participant health is assessed with the following: "Would you say that in general your health is... Select one" And the following choices: "Excellent", "Very good", "Good", "Fair", and "Poor".
Use of other smoking cessation tools | 12 and 26 weeks
  Assessed via self-report. Participants are asked about other smoking cessation tools they have used since the study started. Tools asked about include: cold turkey, apps (other than Pivot), counseling, medications, acupuncture, hypnotherapy, etc. Participants can report other tools not included in the list provided. Outcome reported as the number of participants who have used each other smoking cessation tool.
Change in Alcohol Use Behavior | 12 and 26 weeks
  Assessed via the Alcohol Use Disorders Identification Test-Concise (AUDIT-C) screening questionnaire, 3 items. A score is calculated from a sum of the 3 items. Possible scores on the scale range from 0-12. A score of 0 indicates no alcohol use. Higher scores indicate greater alcohol use behavior, a worse outcome. Scores are compared from baseline to follow-up to determine change in alcohol use behavior.
Change in presence of depressive symptoms | 12 and 26 weeks
  Assessed via the Center of Epidemiological Studies Depression Scale (CES-D) screening questionnaire, 10 items. A score is calculated from a sum of the 10 items. Possible scores on the scale range from 0-30. Higher scores indicate greater severity of depressive symptoms, a worse outcome. Scores are compared from baseline to follow-up to determine change in presence of depressive symptoms.
Living environment relating to nicotine product use and cigarette smoking | 12 and 26 weeks
  Assessed via participant self-report of living with other adults who uses nicotine products other than cigarettes and/or smokes. Participants asked: "Of the adults you live with, how many smoke cigarettes?" and "Of the adults you live with, how many use nicotine products other than cigarettes?". Outcome unit of measure = number of adults.
Living/relationship environment relating to nicotine product use and cigarette smoking | 12 and 26 weeks
  Assessed via participant self-report of living with a romantic partner who uses nicotine products other than cigarettes and/or smokes. Participants asked: "Do you live with a romantic partner who smokes cigarettes?" (yes/no) and "Do you live with a romantic partner who uses nicotine products other than cigarettes?" (yes/no). Outcomes measure reported as number of participants who live with a romantic partner that smokes, and number that live with a romantic partner that uses nicotine products other than cigarettes (participants that answer yes to these questions).
Social environment relating to nicotine product use and cigarette smoking | 12 and 26 weeks
  Assessed via participant self-report of the number of their close friends who use nicotine products other than cigarettes and/or smoke. Participants asked: "How many of your close friends smoke cigarettes?" and "How many of your close friends use nicotine products other than cigarettes?". Outcome unit of measure = number of close friends.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Marler, MD, Principal Investigator — Pivot Health Technologies Inc.
Locations (1):
- Pivot Health Technologies, Inc., San Carlos, California, United States